CLINICAL TRIAL: NCT04734093
Title: Sonographic Signs of Gouty Arthritis in a Cohort of Egyptian Patients: a Cross Sectional Multicenter Study
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Other Study IDs: 21130
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Sonographic Signs of Gouty Arthritis in Diagnosed and Suspected Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Sohag university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Minia university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Assuit university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Kasr Elini recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Tanta university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Monofia university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Aswan university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis
- Ain shams university recruited patients
  Interventions: Diagnostic Test: Evaluation of sonographic signs of gouty arthritis

INTERVENTIONS:
Diagnostic Test: Evaluation of sonographic signs of gouty arthritis — the EULAR scanning protocol for the knee and 1st MTP will be considered [2]. Further, scanning of the double contour sign over the femur condyles anteriorly and posteriorly in sagittal planes will be assessed. Examination of erosions, tophus, double contour, effusion, and echogenic foci will be recorded.

SUMMARY:
The study is a cross sectional observational multicenter study. It is established in collaboration with the Egyptian college of rheumatology study group (ECRsg). It is conditioned that all the study participants had either mono- or oligo-arthritis with effusion of the knee or the first metatarsophalangeal (MTP) joint in patients with a known history of gout or at high risk. Patients with any known chronic arthritis, comprising rheumatoid arthritis, Sjogren's syndrome, systemic lupus erythematosus, scleroderma, neuropathic arthritis, seronegative spondyloarthropathy, will be excluded from the study. None of the participants had a history of intra-articular injection or aspiration in the scanned joints for 3 months prior to the inclusion in the study. The sonographers will be blinded for clinical data and the EULAR scanning protocol for the knee and 1st MTP will be considered [2]. Further, scanning of the double contour sign over the femur condyles anteriorly and posteriorly in sagittal planes will be assessed. All the sonographers in the study had an experience between 5 and 10 years in the field of musculoskeletal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* mono- or oligo-arthritis with effusion of the knee or the first metatarsophalangeal
* patients with a known history of gout or at high risk

Exclusion Criteria:

* Patients with any known chronic arthritis, comprising rheumatoid arthritis, Sjoegren's syndrome, systemic lupus erythematosus, scleroderma, neuropathic arthritis, seronegative spondyloarthropathy
* History of intra-articular injection in the last 3 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be collected from several university clinics all over Egypt. All are aged 40 or more with a history of definite gouty arthritis or at high risk and they have active arthritis of at least one joint.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Sonographic signs of gouty arthritis in the knee or 1st MTP joint | at baseline
  Erosions, effusion, echogenic foci, and tophus using OMERACT definitions of sonographic signs of gouty arthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Elsaman, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No